CLINICAL TRIAL: NCT07327957
Title: The Effect of Vibration and Breathing Exercises Applied Before Chest Tube Removal on Pain and Anxiety: A Randomized Controlled Trial
Brief Title: Effects of Vibration and Breathing Exercises on Pain and Anxiety During Chest Tube Removal
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gamze BULUT (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor-Investigator, Gamze BULUT, Research Assistant, Department of Surgical Nursing, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CTT-VIBREATH-RCT-ATAU-2025
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain; Anxiety; Thoracic Drainage
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders | interventions — Vibration; Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibration and Breathing Exercise Group (Experimental): Participants in this group will receive a combined non-pharmacological intervention consisting of vibration application and guided breathing exercises prior to chest tube removal. The vibration will be applied using a portable vibration device to the area proximal to the chest tube insertion site for a standardized duration. Breathing exercises will be performed under the guidance of the researcher and will include slow, deep, and diaphragmatic breathing techniques aimed at promoting relaxation. All interventions will be administered in addition to routine clinical care.
  Interventions: Other: Vibration and Breathing Exercises
- Control Group (Standard Care) (No Intervention): Participants in the control group will receive routine clinical care according to standard hospital protocols prior to chest tube removal. No additional non-pharmacological interventions, including vibration or breathing exercises, will be applied before the procedure.

INTERVENTIONS:
Other: Vibration and Breathing Exercises — Participants assigned to the intervention group will receive a combined non-pharmacological intervention consisting of vibration application and guided breathing exercises prior to chest tube removal. Vibration will be applied using a portable vibration device placed on the skin near the chest tube insertion site for a standardized duration. The application will be performed while the patient is in a comfortable position.
  Following the vibration application, participants will be guided through structured breathing exercises, including slow, deep, diaphragmatic, and pursed-lip breathing techniques. These exercises will be conducted by the researcher in a calm and quiet environment to promote relaxation. The combined intervention will be administered in addition to routine clinical care and completed before the chest tube removal procedure.
  Arms: Vibration and Breathing Exercise Group

SUMMARY:
Removing a chest tube is a common procedure after chest surgery, but it can cause significant pain and anxiety for patients. Although medications can help reduce these symptoms, they may have side effects and are not always sufficient. Therefore, simple and safe non-drug methods are increasingly used to improve patient comfort.

This randomized controlled study aims to examine the effects of vibration and breathing exercises applied before chest tube removal on patients' pain and anxiety levels. Adult patients with a chest tube will be randomly assigned to one of three groups: a vibration group, a breathing exercise group, or a control group receiving standard care. Pain and anxiety levels will be measured before the procedure and after chest tube removal using validated scales.

The findings of this study are expected to show whether vibration and breathing exercises are effective in reducing pain and anxiety during chest tube removal. If effective, these methods may offer nurses an easy, low-cost, and safe way to improve patient comfort and support evidence-based nursing care.

DETAILED DESCRIPTION:
Chest tube removal is a necessary clinical procedure following thoracic surgery, but it is frequently associated with acute pain and heightened anxiety. These symptoms may negatively affect patient comfort, cooperation, and recovery. While pharmacological interventions are commonly used to manage procedure-related pain and anxiety, concerns regarding side effects and limited effectiveness have increased interest in non-pharmacological approaches within nursing care.

This randomized controlled study is designed to evaluate the effectiveness of vibration and breathing exercises applied prior to chest tube removal on pain and anxiety levels. Eligible adult patients hospitalized in a thoracic surgery unit and scheduled for chest tube removal will be randomly assigned to one of three groups: a vibration group, a breathing exercise group, or a control group receiving routine care. Randomization will be performed using a web-based randomization tool to ensure equal allocation.

In the vibration group, a portable vibration device will be applied to the area proximal to the chest tube insertion site for a standardized duration before the removal procedure. In the breathing exercise group, participants will be guided through structured breathing exercises designed to promote relaxation and diaphragmatic breathing. The control group will receive standard clinical care without any additional non-pharmacological intervention.

Pain intensity and anxiety levels will be assessed at two time points: prior to the chest tube removal procedure and shortly after the procedure. Validated measurement tools will be used to ensure reliability of the findings. Data will be analyzed to compare changes in pain and anxiety levels within and between groups.

The results of this study are expected to provide evidence regarding the use of vibration and breathing exercises as simple, safe, and cost-effective nursing interventions to reduce pain and anxiety associated with chest tube removal. These findings may contribute to the development of evidence-based, non-pharmacological strategies in clinical nursing practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years and older
* Hospitalized patients with an indwelling chest tube scheduled for removal
* First-time chest tube placement
* Conscious, oriented, and cooperative
* Able to understand and communicate in Turkish
* Hemodynamically stable at the time of chest tube removal
* No use of analgesic or sedative medications within 4 hours prior to the procedure
* Willing and able to provide written informed consent

Exclusion Criteria:

* History of any cognitive or psychiatric disorder
* Previous experience with chest tube placement
* Requirement for mechanical ventilation or endotracheal intubation
* Presence of chronic pain or regular use of analgesic medications
* Use of analgesic or sedative medications immediately before chest tube removal
* Unstable clinical condition at the time of the procedure
* Refusal or inability to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Assessed immediately before chest tube removal and 10 minutes after the procedure.
  Pain intensity associated with chest tube removal will be assessed using the Visual Analog Scale (VAS), a validated 10-cm scale ranging from 0 (no pain) to 10 (worst imaginable pain). Participants will self-report their pain level.

SECONDARY OUTCOMES:
Anxiety Level | Assessed immediately before chest tube removal and 10 minutes after the procedure.
  Anxiety levels will be measured using the State Anxiety Inventory (State-Trait Anxiety Inventory - State subscale), a validated self-report questionnaire designed to assess situational anxiety. Higher scores indicate higher levels of anxiety.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The data collected in this study include sensitive health information, and sharing IPD may pose a risk to participant confidentiality and privacy. In addition, the informed consent obtained from participants does not include permission for data sharing beyond the research team. Therefore, IPD will be used solely for the purposes of this study and related scientific